CLINICAL TRIAL: NCT05206682
Title: Comparison of the Therapeutic Effects of Vaginal Repair With Leuprorelin and Vaginal Repair in the Treatment of Cesarean Section Scar Defect
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XH-21-013
Record Dates: First submitted 2022-01-11; First posted 2022-01-25 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-02

CONDITIONS: Cesarean Section; Dehiscence
Keywords: Cesarean Section Scar Defect; Zoladex; vaginal repair
MeSH Terms: interventions — Leuprolide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaginal Repair with Leuprorelin (Experimental): CSD patients were treated with vaginal repair of CSD in combination with Leuprorelin . In the group of Vaginal Repair With Leuprorelin, the patients will get 3 times of Leuprorelin per 4 weeks perioperation. The detailed procedure of Vaginal Repair has been described in our previous study.
  Interventions: Drug: Leuprorelin
- Vaginal Repair without Leuprorelin (No Intervention): The detailed procedure of Vaginal Repair has been described in our previous study.

INTERVENTIONS:
Drug: Leuprorelin — Leuprorelin will be used to postpone period after vaginal repair.
  Arms: Vaginal Repair with Leuprorelin

SUMMARY:
GnRH-a will be used to postpone period after vaginal repair for Cesarean Section Scar Defect（CSD） patients with adenomyosis which will be compared with CSD patients with adenomyosis who receive transvaginal surgery without GnRH-a, whether delayed period improving the CSD prognosis will be assessed.

DETAILED DESCRIPTION:
Women with CSD complicated with adenomyosis will be enrolled in this study. They all will receive vaginal excision and suture of CSD and will be required to undergo examinations at 6-months after surgery.

Interventioned group will be subcutaneous injected of Leuprorelin to postpone period after vaginal repair. It is be assumed that temporary menopause could improve inner conditions of uterus, there would be less local inflammation reaction which would be beneficial to the scar healed.

ELIGIBILITY:
Inclusion Criteria:

1. Clearly diagnosed with CSD complicated with adenomyosis
2. Experiencing clinical features of abnormal uterine bleeding, prolonged menstrual flow (the duration of menstruation is more than 10 days).
3. The thickness of the remaining muscular layer of CSD was less than 3 mm.
4. Normal range of blood sugar and insulin
5. No serious medical problems (important viscera function in the normal range).
6. uterine fibroids no more than 5cm
7. Sign the informed consent.

Exclusion Criteria:

1. Indefinite diagnosis.
2. Malignant tumors.
3. With severe medical problems (severe liver disease, kidney disease, respiratory diseases, heart disease or uncontrolled diabetes, epilepsy, etc., dysfunction of important organs).
4. Pregnant.
5. Mental diseases.
6. Allergy to the any ingredients of Leuprorelin
7. Unwilling to comply with the research plan.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
thickness of the remaining muscular layer (TRM) (mm) | 12 weeks after vaginal repair of CSD
  The thickness of the remaining muscular layer is measured by magnetic resonance imaging (MRI)
Duration of menstruation (day) | 12 weeks after vaginal repair of CSD
  Duration of menstruation (day)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiaotong University xinhua hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No